CLINICAL TRIAL: NCT01361412
Title: An Optional Research Study to Identify Potential Biomarkers of Response to Peptide Immunotherapy for Ragweed Allergy in Subjects Already Enrolled in Clinical Study TR002
Brief Title: Identification of Potential Biomarkers of Response to Peptide Immunotherapy for Ragweed Allergy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Circassia Limited (Industry)
Collaborators: Adiga Life Sciences, Inc. (Industry); Cetero Research, San Antonio (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double
Other Study IDs: TR002A
Record Dates: First submitted 2011-05-24; First posted 2011-05-26 (Estimated); Last update posted 2011-10-07 (Estimated); Status verified 2011-10

CONDITIONS: Ragweed Allergy
Keywords: ragweed allergy; immunotherapy

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (5):
- ToleroMune Ragweed 4 (Experimental)
  Interventions: Biological: ToleroMune Ragweed
- ToleroMune Ragweed Regimen 3 (Experimental)
  Interventions: Biological: ToleroMune Ragweed
- ToleroMune Ragweed Regimen 2 (Experimental)
  Interventions: Biological: ToleroMune Ragweed
- Placebo (Placebo Comparator): Placebo
  Interventions: Biological: Placebo
- ToleroMune Ragweed Regimen 1 (Experimental)
  Interventions: Biological: ToleroMune Ragweed

INTERVENTIONS:
Biological: ToleroMune Ragweed — Intradermal administration 1x8 administrations, 2 weeks apart
  Arms: ToleroMune Ragweed 4; ToleroMune Ragweed Regimen 1; ToleroMune Ragweed Regimen 2; ToleroMune Ragweed Regimen 3
Biological: Placebo — Intradermal injection 1x8 administrations, 2 weeks apart
  Arms: Placebo

SUMMARY:
The aim of the study is to identify changes in potential biomarkers after peptide immunotherapy for that may subsequently be developed as biomarkers that correlate with clinical efficacy.

ELIGIBILITY:
Inclusion Criteria:

* Enrolled in study TR002 but have not yet commenced dosing

Exclusion Criteria:

* None; no criteria additional to TR002 exclusion criteria are applicable to this study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2011-03; Primary Completion 2011-09 (Actual); Study Completion 2011-09 (Actual)

PRIMARY OUTCOMES:
Identification of potential plasma biomarkers of response to peptide immunotherapy | 6 months after start of dosing
  Blood samples derived from the study will be submitted for proteomics analyses aimed at the identification of one or more plasma proteins whose concentration over the course of the study varies in relation to the treatment administered. The outcome will be determined on the basis of measurements from samples collected over a period commencing prior to treatment and ending 6 months following treatmen

CONTACTS AND LOCATIONS:
Overall Officials: Deepen Patel, MD, CCFP, Principal Investigator — Cetero Research, San Antonio
Locations (1):
- Cetero Research, Mississauga, Ontario, Canada